CLINICAL TRIAL: NCT07335692
Title: Dynamical Electrophysiology and Neuropathology in Lewy's Bodies Disease
Acronym: DYNAPATH-LB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9691
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lewy Body Disease
Keywords: Lewy Body Disease; Neurodegenerative disorder
MeSH Terms: conditions — Lewy Body Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lewy body disease (LBD) is a neurodegenerative disorder that causes cognitive and behavioral problems. However, it is difficult to diagnose, and its pathophysiology is still not fully understood. The usual diagnostic criteria for LBD have excellent specificity but poor sensitivity. In particular, we lack paraclinical tests that can make a significant contribution. LBD patients may exhibit abnormalities in brain activity dynamics, which can be detected by EEG and may be linked to neuronal dysfunctions specific to the disease. The objective of this study is twofold: first, to assess the validity of this observation, that is, to confirm that the observed phenomenon is indeed linked to the pathophysiology of LBD, and second, to clarify the nature of these abnormalities by exploring the brain dynamics of LBD patients in greater detail.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥18 years old).
* Subject who participated in the Alpha-Lewy-MA cohort and underwent RT-QuIC analysis.
* Subject who underwent a standard EEG examination at HUS between January 1, 2012, and January 1, 2020.

Exclusion Criteria:

- Subject who expressed opposition to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (≥18 years old) who participated in the Alpha-Lewy-MA cohort and underwent RT-QuIC analysis and underwent a standard EEG examination at HUS between January 1, 2012, and January 1, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Parameter θ of dynamic fluidity of brain activity | Up to 12 months
  Parameter θ of dynamic fluidity of brain activity (quantifying the system's ability to move away from its current configuration)
  θ is used to measure something specific in the brain: how flexible its activity is.
  Quantifying the system's ability to move away from its current configuration:
  * In plain words, θ tells us how much the brain can change from its current state.
  * High θ → brain is very flexible, can switch between states easily.
  * Low θ → brain is rigid, stays in the same pattern longer.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de psychiatrie de la personne âgée - CHU de Strasbourg - France, Strasbourg, France